CLINICAL TRIAL: NCT03974971
Title: Blastic Plasmacytoid Dendritic Cell Neoplasm in Korean Population: A Multicenter Study
Brief Title: Blastic Plasmacytoid Dendritic Cell Neoplasm in Korean Population.
Acronym: KBPDCN
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Kim, Seok Jin, Principal Investigator, Samsung Medical Center
Other Study IDs: 2019-02-035
Record Dates: First submitted 2019-05-22; First posted 2019-06-05 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Blastic Plasmacytoid Dendritic Cell Neoplasm
MeSH Terms: conditions — Blastic Plasmacytoid Dendritic Cell Neoplasm

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BPDCN diagnosis group: By review medical records Enroll patients diagnosed with BPDCN from January 1, 2000 to October 31, 2018

SUMMARY:
Retrospective study , To analyze the clinical features and treatment outcomes in Korean blastic plasmacytoid dendritic cell neoplasm.

DETAILED DESCRIPTION:
Blastic plasmacytoid dendritic cell neoplasm (BPDCN), with a synonym of blastic NK-cell lymphoma, agranular CD4+ natural killer cell leukaemia, blastic natural killer leukaemia/lymphoma, and agranular CD4+CD56+ haematodermic neoplasm/tumour, has been classified under "acute myeloid leukemia (AML) and related precursor neoplasms" since 2008 according to the World Health Organization (WHO) classification and among "myeloid neoplasm and acute leukemia" following 2016 revision of WHO classification. The plasmacytoid dendritic cells originates professional type I interferon-producing cells or plasmacytoid monocytes. Therefore, the prerequisite for diagnosis of BPDCN is the CD4+ and CD 56+ co-expression without common lymphoid or myeloid lineage markers1,2. This rare type of malignancy affecting predominantly elderly man, is reported to comprise 0.44% of hematologic malignancy3 and 0.7% of cutaneous lymphomas4, and the leukemic presentation or transformation is observed at initial presentation or even in the course of disease progression5.

Skin in¬volvement is a predominant clinical feature of BPDCN ranging in appearance from small bruise-like areas to patches, nodules, and ulcerated masses, but lymphadenopathy, splenomegaly, hepatomegaly are also commonly observed. There is no definite treatment guideline for BPDCN. Retrospective studies including acute myeloid leukemia (AML) or acute lymphoblastic leukemia (ALL)/lymphoma-like chemotherapy for management of BPDCN reported 53-89% of high complete remission rates but an eventual very poor overall survival of 12-23 months, with a preponderance of ALL/lymphoma- over AML-like treatment5. Recently, targeted therapy with SL401, an IL-3 fusion protein which binds to CD123, is promising and the results of the clinical trial will be unveiled in the near future6.

Although several retrospective and small case series has been published so far7,8, there is still no multicenter study on BPDCN classified after 2008 WHO classification in Asian population. This study aims to retrospectively collect data of BPDCN patients from centers participating the Consortium for improving survival of lymphoma (CISL) and analyze the clinical features and treatment outcomes in this rare type of hematologic malignancy.

ELIGIBILITY:
<Inclusion Criteria>

1. Patients ≥ 18 years
2. Pathologically confirmed diagnosis by tissue or bone marrow at each center with

   * Blastic plasmacytoid dendritic cell neoplasm
   * Blastic NK-cell lymphoma
   * Agranular CD4+ natural killer cell leukaemia
   * Blastic natural killer leukaemia/lymphoma
   * Agranular CD4+CD56+ haematodermic neoplasm/tumour
3. Antigen expression of CD4 and/or CD56 coupled with at least one plasmacytoid dendritic cell-associated antigen among CD123, TCL1, CD2AP and BDCA2/CD303

<Exclusion Criteria>

1. Acute myeloid leukemia
2. Acute lymphoblastic leukemia
3. Mixed phenotype acute leukemia
4. Any type of B- or T-/NK/T-cell lymphomas
5. Expression of lineage-specific markers for B cells (CD20, CD79a) T cells (CD3) Myeloid cells (myeloperoxidase) Monocytes (CD11c, CD163, lysozyme). CD34

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study is a retrospective study, in which patients with patients diagnosed with SCC tumors can participate, and patients who meet the selection criteria will be eligible. The purpose of this study is explorative and descriptive, and it is impossible to calculate the statistical background. Therefore, it is estimated that more than 40 patients are diagnosed with the disease in Korea so far.
Sampling Method: Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Overall Survival Rate | from the date of the IRB approval until June 30, 2019
  From the date of diagnosis to the date of death, or from the date of diagnosis to the last follow-up date.

SECONDARY OUTCOMES:
Therapeutic Response Rate | from the date of the IRB approval until June 30, 2019
  Therapeutic response analysis is based on the evaluation of the response of common leukemia and lymphoma
Disease-free Survival Rate | from the date of the IRB approval until June 30, 2019
  the time from the treatment start date until the patient recurs.
Number of Factors affecting overall survival | from the date of the IRB approval until June 30, 2019
  multivariate analysis of age, ECOG, Involving organs, Response to treatment, Treatment, Autologous transplantation/Allogeneic transplantation affecting overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Seokjin Kim, M.D., PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung medical center, Seoul, Gang Nam, South Korea

IPD SHARING:
Plan to Share IPD: No